CLINICAL TRIAL: NCT05466214
Title: Systematic Efficacy Replication Study of Conjoint Behavioral Consultation in Elementary Schools
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American Institutes for Research (Other)
Collaborators: Wisconsin Center for Education Research (Unknown); University of Nebraska College of Education and Human Sciences (Unknown)
Responsible Party: Principal Investigator, Elizabeth Spier, Principal Researcher, American Institutes for Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Systematic Efficacy CBC 2021
Record Dates: First submitted 2022-04-05; First posted 2022-07-20 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Emotional Disturbances
MeSH Terms: conditions — Affective Symptoms

STUDY DESIGN:
Intervention Model Description: Conjoint Behavioral Consultation (CBC) is an indirect consultation process focused on ameliorating problematic behaviors associated with severe emotional disturbance through structured, data-based problem solving and collaborative, consistent implementation of evidence-based interventions across home and school settings, while simultaneously enhancing family-school partnerships.. In CBC, problems are identified, defined, analyzed, and treated through strengths-based, mutual, collaborative interactions between parents and teachers with the support of a consultant. Through CBC, parents and teachers are taught evidence-based procedures to address behavior problems in their respective settings. Parents and teachers assume complementary roles and shared responsibility for identifying student goals and addressing challenging behaviors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBC Treatment Group (Experimental): For this group, school staff who work with families and teachers to address student emotional and behavioral concerns will use the CBC model to do so.
  Interventions: Behavioral: Conjoint Behavioral Consultation (CBC)
- Control Group (No Intervention): For this group, school staff who work with families and teachers to address student emotional and behavioral concerns will engage in business as usual.

INTERVENTIONS:
Behavioral: Conjoint Behavioral Consultation (CBC) — Within the treatment group, CBC will be integrated into how a school-based specialist works with families and teachers of children with or at risk of severe emotional disturbance.
  Other Names: Teachers and Parents as Partners (TAPP)
  Arms: CBC Treatment Group

SUMMARY:
The purpose of this project is to conduct an impact evaluation of the Conjoint Behavioral Consulting (CBC) intervention under real-world conditions as an IES Efficacy Replication trial. CBC is a family-school partnership intervention proven efficacious for children with serious emotional and behavior problems. The investigation will conduct a systematic efficacy replication of CBC to identify important process and context variables in need of attention prior to a CBC effectiveness study. School-based specialists (SBSs) will implement CBC and will be responsible for working directly with parents and teachers who have a student with or at risk for severe emotional disturbance, with more implementation support (i.e., non-routine conditions) than would be expected under routine conditions to ensure adequate fidelity of implementation. The research questions examine the impact of CBC, when implemented by SBSs, on student, parent, and teacher outcomes, as well its effect on mediational pathways. In addition, the research team will gather stakeholder feedback in focus groups to provide information about factors that stakeholders perceive as impeding or promoting CBC adoption, implementation, and sustainability.

DETAILED DESCRIPTION:
Sixty schools will be recruited for this impact evaluation (20 from Madison Metropolitan School District, and 40 from Milwaukee Public Schools). The population for this evaluation will consist of the 12 children from grades k-4 in each participating school who demonstrate the highest levels of behavioral and/or emotional difficulties in school, based on teacher ratings on the BASC3-BESS screening (and whose families consent to participate in the evaluation). The total population for this evaluation will include 720 students. Baseline will take place at the beginning of the intervention school year, outcome 1 at the end of the intervention school year, and outcome 2 at the end of the subsequent school year. At all three timepoints, the research team will gather parent questionnaires (covering competence in problem solving, parenting strategies, parent-teacher relationships, and their child's social and behavioral functioning), teacher questionnaires in relation to each study child (covering the parent-teacher relationship, teacher competence in problem solving, and the student's social and behavioral functioning), direct observations of teacher and student behavior in the classroom, and student records related to discipline.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in kindergarten, Grade 1, Grade 2, Grade 3, or Grade 4 at recruitment
* Among the 12 students with the highest risk score on the Behavioral and Emotional Screening System 3 Behavioral and Emotional Screening System (BASC3-BESS) in the above grade span in their school (among those with parental consent for screening).

Exclusion Criteria: None

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Child Externalizing Problems, Parent Report, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in children's norm-referenced t-scores on the Externalizing Problems subscale of the Behavior Assessment System for Children, Third Edition, parent report version.
Child Externalizing Problems, Teacher Report, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in children's norm-referenced t-scores on the Externalizing Problems subscale of the Behavior Assessment System for Children, Third Edition, teacher report version.
Child Externalizing Problems, Parent Report, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in children's norm-referenced t-scores on the Externalizing Problems subscale of the Behavior Assessment System for Children, Third Edition, parent report version.
Child Externalizing Problems, Techer Report, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in children's norm-referenced t-scores on the Externalizing Problems subscale of the Behavior Assessment System for Children, Third Edition, teacher report version.
Child Internalizing Problems, Parent Report, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in children's norm-referenced t-scores on the Internalizing Problems subscale of the Behavior Assessment System for Children, Third Edition, parent report version.
Child Internalizing Problems, Teacher Report, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in children's norm-referenced t-scores on the Internalizing Problems subscale of the Behavior Assessment System for Children, Third Edition, teacher report version.
Child Internalizing Problems, Parent Report, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in children's norm-referenced t-scores on the Internalizing Problems subscale of the Behavior Assessment System for Children, Third Edition, parent report version.
Child Internalizing Problems, Teacher Report, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in children's norm-referenced t-scores on the Internalizing Problems subscale of the Behavior Assessment System for Children, Third Edition, teacher report version.
Child Behavioral Symptoms, Parent Report, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in children's norm-referenced t-scores on the Behavioral Symptoms subscale of the Behavior Assessment System for Children, Third Edition, parent report version.
Child Behavioral Symptoms, Teacher Report, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in children's norm-referenced t-scores on the Behavioral Symptoms subscale of the Behavior Assessment System for Children, Third Edition, teacher report version.
Child Behavioral Symptoms, Parent Report, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in children's norm-referenced t-scores on the Behavioral Symptoms subscale of the Behavior Assessment System for Children, Third Edition, parent report version.
Child Behavioral Symptoms, Teacher Report, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in children's norm-referenced t-scores on the Behavioral Symptoms subscale of the Behavior Assessment System for Children, Third Edition, teacher report version.
Child Adaptive Skills, Parent Report, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in children's norm-referenced t-scores on the Adaptive Skills subscale of the Behavior Assessment System for Children, Third Edition, parent report version.
Child Adaptive Skills, Teacher Report, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in children's norm-referenced t-scores on the Adaptive Skills subscale of the Behavior Assessment System for Children, Third Edition, teacher report version.
Child Adaptive Skills, Parent Report, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in children's norm-referenced t-scores on the Adaptive Skills subscale of the Behavior Assessment System for Children, Third Edition, parent report version.
Child Adaptive Skills, Teacher Report, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in children's norm-referenced t-scores on the Adaptive Skills subscale of the Behavior Assessment System for Children, Third Edition, teacher report version.
Child School Problems, Teacher Report, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in children's norm-referenced t-scores on the School Problems subscale of the Behavior Assessment System for Children, Third Edition, teacher report version.
Child School Problems, Teacher Report, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in children's norm-referenced t-scores on the School Problems subscale of the Behavior Assessment System for Children, Third Edition, teacher report version.
Child Social Skills, Parent Report, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in children's norm-referenced t-scores on the Social Skills subscale of the Social Skills Improvement System Rating Scales, parent report version.
Child Social Skills, Teacher Report, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in children's norm-referenced t-scores on the Social Skills subscale of the Social Skills Improvement System Rating Scales, teacher report version.
Child Social Skills, Parent Report, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in children's norm-referenced t-scores on the Social Skills subscale of the Social Skills Improvement System Rating Scales, parent report version.
Child Social Skills, Teacher Report, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in children's norm-referenced t-scores on the Social Skills subscale of the Social Skills Improvement System Rating Scales, teacher report version.
Child Problem Behaviors, Parent Report, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in children's norm-referenced t-scores on the Problem Behaviors subscale of the Social Skills Improvement System Rating Scales, parent report version.
Child Problem Behaviors, Teacher Report, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in children's norm-referenced t-scores on the Problem Behaviors subscale of the Social Skills Improvement System Rating Scales, teacher report version.
Child Problem Behaviors, Parent Report, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in children's norm-referenced t-scores on the Problem Behaviors subscale of the Social Skills Improvement System Rating Scales, parent report version.
Child Problem Behaviors, Teacher Report, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in children's norm-referenced t-scores on the Problem Behaviors subscale of the Social Skills Improvement System Rating Scales, teacher report version.
Child Autism Behaviors, Parent Report, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in children's norm-referenced t-scores on the Autism Behaviors subscale of the Social Skills Improvement System Rating Scales, parent report version.
Child Autism Behaviors, Teacher Report, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in children's norm-referenced t-scores on the Autism Behaviors subscale of the Social Skills Improvement System Rating Scales, teacher report version.
Child Autism Behaviors, Parent Report, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in children's norm-referenced t-scores on the Autism Behaviors subscale of the Social Skills Improvement System Rating Scales, parent report version.
Child Autism Behaviors, Teacher Report, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in children's norm-referenced t-scores on the Autism Behaviors subscale of the Social Skills Improvement System Rating Scales, teacher report version.
Parenting Strategies: Consistent Discipline, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for the Consistent Discipline subscale of the Parenting Strategies instrument. Scores are calculated based on the mean rating across 11 items, with possible mean scores ranging from 1-5.
Parenting Strategies: Consistent Discipline, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in score for the Consistent Discipline subscale of the Parenting Strategies instrument. Scores are calculated based on the mean rating across 11 items, with possible mean scores ranging from 1-5.
Parenting Strategies: Parental Acceptance, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for the Parental Acceptance subscale of the Parenting Strategies instrument. Scores are calculated based on the mean rating across 8 items, with possible mean scores ranging from 1-5.
Parenting Strategies: Parental Acceptance, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in score for the Parental Acceptance subscale of the Parenting Strategies instrument. Scores are calculated based on the mean rating across 8 items, with possible mean scores ranging from 1-5.
Parenting Strategies: Positive Reinforcement, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for the Positive Reinforcement subscale of the Parenting Strategies instrument. Scores are calculated based on the mean rating across 12 items, with possible mean scores ranging from 1-5.
Parenting Strategies: Positive Reinforcement, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in score for the Positive Reinforcement subscale of the Parenting Strategies instrument. Scores are calculated based on the mean rating across 12 items, with possible mean scores ranging from 1-5.
Teacher Strategies: Positive Strategies, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for the Positive Strategies subscale of the Teacher Strategies instrument. Scores are calculated based on the mean rating across 22 items, with possible mean scores ranging from 1-5.
Teacher Strategies: Inappropriate Strategies, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for the Inappropriate Strategies subscale of the Teacher Strategies instrument. Scores are calculated based on the mean rating across 9 items, with possible mean scores ranging from 1-5.
Parent-Teacher Relationship: Parent Perspective on Joining, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for the Joining subscale of the Parent-Teacher Relationship Scale II, parent version. Scores are calculated based on the mean rating across 19 items, with possible mean scores ranging from 1-5.
Parent-Teacher Relationship: Teacher Perspective on Joining, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for the Joining subscale of the Parent-Teacher Relationship Scale II, teacher version. Scores are calculated based on the mean rating across 19 items, with possible mean scores ranging from 1-5.
Parent-Teacher Relationship: Parent Perspective on Communication, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for the Communication subscale of the Parent-Teacher Relationship Scale, parent version. Scores are calculated based on the mean rating across 5 items, with possible mean scores ranging from 1-5.
Parent-Teacher Relationship: Teacher Perspective on Communication, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for the Communication subscale of the Parent-Teacher Relationship Scale, teacher version. Scores are calculated based on the mean rating across 5 items, with possible mean scores ranging from 1-5.
Parent Competence in Problem Solving, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for the Parent Competence in Problem Solving Scale. Scores are calculated based on the mean rating across 8 items, with possible mean scores ranging from 1-6.
Teacher Competence in Problem Solving, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for the Teacher Competence in Problem Solving Scale. Scores are calculated based on the mean rating across 8 items, with possible mean scores ranging from 1-6.
Parent Competence in Problem Solving, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in score for the Parent Competence in Problem Solving Scale. Scores are calculated based on the mean rating across 8 items, with possible mean scores ranging from 1-6.
Behavior Watch Student: Inappropriate Motor Activity, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for Inappropriate Motor Activity on the Behavior Watch observation tool, student version. Scores are calculated based on the rate observed for intervals recorded, with a possible score of 0.0-1.0.
Behavior Watch Student: Inappropriate Motor Activity, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in score for Inappropriate Motor Activity on the Behavior Watch observation tool, student version. Scores are calculated based on the rate observed for intervals recorded, with a possible score of 0.0-1.0.
Behavior Watch Student: Off Task, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for Off Task on the Behavior Watch observation tool, student version. Scores are calculated based on the rate observed for intervals recorded, with a possible score of 0.0-1.0.
Behavior Watch Student: Off Task, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in score for Off Task on the Behavior Watch observation tool, student version. Scores are calculated based on the rate observed for intervals recorded, with a possible score of 0.0-1.0.
Behavior Watch Student: On Task, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for On Task on the Behavior Watch observation tool, student version. Scores are calculated based on the rate observed for intervals recorded, with a possible score of 0.0-1.0.
Behavior Watch Student: On Task, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in score for On Task on the Behavior Watch observation tool, student version. Scores are calculated based on the rate observed for intervals recorded, with a possible score of 0.0-1.0.
Behavior Watch Student: Appropriate Interactions, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for Appropriate Interactions on the Behavior Watch observation tool, student version. Scores are calculated based on the rate observed for intervals recorded, with a possible score of 0.0-1.0.
Behavior Watch Student: Appropriate Interactions, Outcome 2 | Baseline/pre-intervention (beginning of school year 1) to end of school year 2 (approximately 19 months)
  Change in score for Appropriate Interactions on the Behavior Watch observation tool, student version. Scores are calculated based on the rate observed for intervals recorded, with a possible score of 0.0-1.0.
Behavior Watch Teacher: Positive Tangible Consequences, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for Positive Tangible Consequences on the Behavior Watch observation tool, teacher version. Scores are calculated based on the rate observed for intervals recorded, with a possible score of 0.0-1.0.
Behavior Watch Teacher: Effective Command, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for Effective Command on the Behavior Watch observation tool, teacher version. Scores are calculated based on the rate observed for intervals recorded, with a possible score of 0.0-1.0.
Behavior Watch Teacher: Positive Attention, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for Positive Attention on the Behavior Watch observation tool, teacher version. Scores are calculated based on the rate observed for intervals recorded, with a possible score of 0.0-1.0.
Behavior Watch Teacher: Use of Reductive Techniques, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for Use of Reductive Techniques on the Behavior Watch observation tool, teacher version. Scores are calculated based on the rate observed for intervals recorded, with a possible score of 0.0-1.0.
Behavior Watch Teacher: Negative Attention, Outcome 1 | Baseline/pre-intervention (beginning of school year 1) to end of school year 1 (approximately 7 months)
  Change in score for Use of Negative Attention on the Behavior Watch observation tool, teacher version. Scores are calculated based on the rate observed for intervals recorded, with a possible score of 0.0-1.0.

CONTACTS AND LOCATIONS:
Overall Officials: Andy Garbacz, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Madison Metropolitan School District, Madison, Wisconsin, United States